CLINICAL TRIAL: NCT01704495
Title: A 6-month, Randomised, Double-blind, Placebo-controlled, Multi-centre, Parallel-group, Phase II Study With an Optional Safety Extension Treatment Period up to 6 Months, to Evaluate the Efficacy, Safety, and Tolerability of 3 Different Doses of AZD5069 Twice Daily as Add-on Treatment to Medium to High Dose Inhaled Corticosteroids (ICS) and Long-acting β2 Agonists (LABA), in Patients With Uncontrolled Persistent Asthma
Brief Title: A Phase II Study to Evaluate the Efficacy, Safety and Tolerability of AZD5069 in Patients With Uncontrolled Persistent Asthma.
Acronym: NIMBUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3551C00001; 2012-001869-33
Record Dates: First submitted 2012-10-09; First posted 2012-10-11 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Uncontrolled Asthma,; Exacerbation,; Safety
MeSH Terms: conditions — Asthma | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- AZD5069 5 mg (Experimental): AZD5069 oral capsules self-administered twice daily
  Interventions: Drug: AZD5069
- AZD5069 15 mg (Experimental): AZD5069 oral capsules self-administered twice daily
  Interventions: Drug: AZD5069
- AZD5069 45 mg (Experimental): AZD5069 oral capsules self-administered twice daily
  Interventions: Drug: AZD5069
- Placebo (Placebo Comparator): Placebo oral capsules self-administered twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5069 — AZD5069 oral capsules self-administered twice daily.
  Arms: AZD5069 15 mg; AZD5069 45 mg; AZD5069 5 mg
Drug: Placebo — Placebo oral capsules self-administered twice daily.
  Arms: Placebo

SUMMARY:
The purpose is to Evaluate the Efficacy, Safety, and Tolerability of 3 Different Doses of AZD5069 Twice Daily as Add-on Treatment to Medium to High Dose Inhaled Corticosteroids (ICS) and Long-acting β2 Agonists (LABA), in Patients with Uncontrolled Persistent Asthma

DETAILED DESCRIPTION:
A 6-month, Randomised, Double-blind, Placebo-controlled, Multi-centre, Parallel-group, Phase II Study with an Optional Safety Extension Treatment Period up to 6 months, to Evaluate the Efficacy, Safety, and Tolerability of 3 Different Doses of AZD5069 Twice Daily as Add-on Treatment to Medium to High Dose Inhaled Corticosteroids (ICS) and Long-acting β2 Agonists (LABA), in Patients with Uncontrolled Persistent Asthma

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and above. Females of childbearing potential must use a highly effective contraceptive method plus a condom by their male partner.
* Diagnosis of asthma for at least 12 months (GINA 2011)
* Uncontrolled persistent asthma, despite treatment with medium to high dose ICS and LABA, and with a history of exacerbations during the last year
* Morning prebronchodilator FEV1 of ≥30% and ≤85% predicted normal at enrolment
* Daily use of medium or high dose ICS (≥fluticasone 500 µg or the equivalent daily)

Exclusion Criteria:

* Any clinically significant disease or disorder (including any chronic lower respiratory disease other than asthma) that may put the patient at risk or influence study results
* Patients with recurrent, latent, or chronic infections
* Active tuberculosis or latent tuberculosis without completion of an appropriate course of treatment or prophylactic treatment
* Significant lower respiratory tract infection not resolved within 30 days prior to enrolment
* Current smoker or smoking history of more than 20 pack years

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Larsson, MEDICAL SCIENCE DIRECTOR, Study Director — AZ Mondal R&D, Sweden
Locations (96):
- Bulgaria (8):
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Razgrad
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Vidin
- Canada (6):
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint Romuald, Quebec
- Czechia (8):
  - Research Site, Brno
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Kutná Hora
  - Research Site, Mělník
  - Research Site, Prague
  - Research Site, Strakonice
  - Research Site, Tábor
- Germany (5):
  - Research Site, Berlin
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, München
- Hungary (14):
  - Research Site, Aszód
  - Research Site, Baja
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Gyula
  - Research Site, Komárom
  - Research Site, Makó
  - Research Site, Monor
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Szombathely
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Giżycko
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Skierniewice
  - Research Site, Tarnów
  - Research Site, Wroclaw
  - Research Site, Żnin
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Deva
  - Research Site, Iași
- Russia (7):
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Vladikavkaz
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (11):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Poprad
  - Research Site, Spišská Nová Ves
  - Research Site, Šurany
  - Research Site, Topoľčany
  - Research Site, Trenčín
  - Research Site, Zvolen
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eManzimtoti
  - Research Site, eMkhomazi
  - Research Site, Pretoria
- Ukraine (8):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
  - Research Site, Zaporizhzhzya
  - Research Site, Zaporozye
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Dundee
  - Research Site, Liverpool
  - Research Site, London

REFERENCES:
- [Derived] O'Byrne PM, Metev H, Puu M, Richter K, Keen C, Uddin M, Larsson B, Cullberg M, Nair P. Efficacy and safety of a CXCR2 antagonist, AZD5069, in patients with uncontrolled persistent asthma: a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2016 Oct;4(10):797-806. doi: 10.1016/S2213-2600(16)30227-2. Epub 2016 Aug 27. PMID 27574788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 months double-blind study with optional safety extension for up to 6 months, were subjects continued on the treatment they were randomized to. First subject enrolled 27 Nov 2012 Last subject last visit 27 Aug 2014 1146 subjects enrolled in tot of which 506 patients were not randomized since they did not fulfilled all the inclusion conditions.
Pre-assignment Details: 4 weeks run-in period on background therapy prior to randomization.
  The discrepancy in the number of enrolled patients compared to the protocol section (n=1147) is because of a patient was in error reported by a monitor as enrolled when the patient was in effect not enrolled.
Groups:
- AZD5069 45 mg BID; AZD5069 15 mg BID; AZD5069 5 mg BID: AZD5069 oral capsules self-administered twice daily
- Placebo: Placebo oral capsules self-administred twice daily
Period: Subjects Randomized
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Started | 162 | 156 | 160 | 162
Completed | 140 | 141 | 144 | 145
Not Completed | 22 | 15 | 16 | 17
Not completed — Other Reason | 3 | 2 | 3 | 2
Not completed — Discontinuation criteria met | 4 | 2 | 2 | 0
Not completed — Adverse Event | 8 | 2 | 0 | 7
Not completed — Withdrawal by Subject | 5 | 5 | 5 | 5
Not completed — Protocol Violation | 1 | 1 | 2 | 0
Not completed — Eligibility criteria not fulfilled | 1 | 3 | 4 | 3
Period: Optional Safety Extension
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Started | 116 (46 subjects did not enter safety extension) | 121 (35 subjects did not enter safety extension) | 114 (46 subjects did not enter safety extension) | 116 (46 subjects did not enter safety extension)
Completed | 87 | 88 | 83 | 85
Not Completed | 29 | 33 | 31 | 31
Not completed — Adverse Event | 0 | 4 | 0 | 1
Not completed — Other reason | 27 | 29 | 30 | 28
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo | Total
Number analyzed (Participants) | 162 | 156 | 160 | 162 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.6) | 52 (12.7) | 53 (11.5) | 54 (11.1) | 52 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 113 | 104 | 120 | 444
  Male | 55 | 43 | 56 | 42 | 196
FEV1 pre-bronchodilator [Median (Full Range); unit: percentage of predicted normal] | 63.74 [30.11 to 85.41] | 66.35 [29.92 to 113.57] | 65.76 [32.57 to 123.86] | 61.58 [31.13 to 84.86] | 64.93 [29.92 to 123.86]
FEV1 post-bronchodilator [Median (Full Range); unit: percentage of predicted normal] | 74.34 [32.33 to 105.44] | 77.95 [30.38 to 112.83] | 76.31 [34.88 to 112.89] | 72.19 [31.26 to 111.88] | 75.22 [30.38 to 112.89]
Reversibility [Mean (Standard Deviation); unit: percentage change] | 18.73 (20.617) | 16.05 (15.580) | 18.41 (20.574) | 18.45 (16.342) | 17.93 (18.438)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Severe Asthma Exacerbations During 6 Months
Time Frame: From start of treatment up to 6 months
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Exacerbations per 6 month
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 161 | 153 | 156 | 159
Exacerbations per 6 month | 0.31 [0.20 to 0.50] | 0.31 [0.19 to 0.49] | 0.26 [0.16 to 0.42] | 0.20 [0.12 to 0.33]
Statistical Analysis 1: Comparison: AZD5069 45 mg BID vs Placebo; Test type: Superiority or Other; p = 0.119, Poisson regression — 2-sided p-value; Correction for overdispersion made by Pearson chi-square; Risk Ratio (RR) = 1.56, 90% CI 2-sided [0.98 to 2.49] — AZD5069 45 mg BID vs Placebo
Statistical Analysis 2: Comparison: AZD5069 15 mg BID vs Placebo; Test type: Superiority or Other; p = 0.141, Poisson Regression — 2-sided; Correction for overdispersion made by Pearson chi-square; Risk Ratio (RR) = 1.53, 90% CI 2-sided [0.95 to 2.46] — AZD5069 15 mg BID vs Placebo
Statistical Analysis 3: Comparison: AZD5069 5 mg BID vs Placebo; Test type: Superiority or Other; p = 0.397, Poisson Regression — 2-sided; Correction for overdispersion made by Pearson chi-square; Risk Ratio (RR) = 1.29, 90% CI 2-sided [0.79 to 2.11] — AZD5069 5 mg BID vs Placebo

2. Secondary Outcome: Rate of Asthma-specific Hospital Admission/Intensive Care Unit Admissions During 6 Months
Time Frame: From start of treatment up to 6 months
Measure: Least Squares Mean (90% Confidence Interval); unit: Exacerbations per 6 month
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 161 | 153 | 156 | 159
Exacerbations per 6 month | 0.04 [0.01 to 0.14] | 0.02 [0.00 to 0.09] | 0.02 [0.02 to 0.09] | 0.02 [0.01 to 0.09]

3. Secondary Outcome: Total Number of Days of Asthma-specific Hospital Admission/Intensive Care Unit Admissions
Time Frame: From start of treatment up to 6 months
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 161 | 153 | 156 | 159
Days | 0.54 [0.26 to 1.12] | 0.82 [0.38 to 1.77] | 0.00 [0.00 to 0.01] | 0.08 [0.03 to 0.23]

4. Secondary Outcome: Total Number of Days on Oral Cortecosteroids, Due to a Worsening of Asthma Symptoms
Time Frame: From start of treatment up to 6 months
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 161 | 153 | 156 | 159
Days | 2.38 [1.33 to 4.26] | 2.43 [1.33 to 4.45] | 2.74 [1.42 to 5.29] | 1.55 [0.80 to 3.00]

5. Secondary Outcome: Change From Baseline to 2 Weeks Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at two weeks are included in the analysis
Time Frame: Baseline (Day 0) and 2 weeks after Day 0
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 155 | 145 | 149 | 155
L | 0.13 [0.06 to 0.20] | 0.07 [0.00 to 0.14] | 0.09 [0.02 to 0.16] | 0.12 [0.05 to 0.19]

6. Secondary Outcome: Change From Baseline to 1 Month Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at one month are included in the analysis
Time Frame: Baseline (Day 0) and 1 month after Day 0
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 153 | 146 | 146 | 153
L | 0.14 [0.07 to 0.21] | 0.08 [0.01 to 0.16] | 0.09 [0.02 to 0.16] | 0.09 [0.02 to 0.16]

7. Secondary Outcome: Change From Baseline to 2 Months Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at two months are included in the analysis
Time Frame: Baseline (Day 0) and 2 months after Day 0
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 150 | 143 | 145 | 150
L | 0.13 [0.06 to 0.20] | 0.08 [0.01 to 0.16] | 0.07 [-0.01 to 0.14] | 0.12 [0.05 to 0.19]

8. Secondary Outcome: Change From Baseline to 3 Months Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at three months are included in the analysis
Time Frame: Baseline (Day 0) and 3 months after Day 0
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 146 | 142 | 145 | 149
L | 0.10 [0.03 to 0.18] | 0.11 [0.04 to 0.18] | 0.06 [-0.02 to 0.13] | 0.06 [-0.01 to 0.13]

9. Secondary Outcome: Change From Baseline to 4 Months Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at four months are included in the analysis
Time Frame: Baseline (Day 0) and 4 months after Day 0
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 148 | 142 | 146 | 148
L | 0.17 [0.09 to 0.24] | 0.17 [0.09 to 0.24] | 0.14 [0.06 to 0.21] | 0.16 [0.08 to 0.23]

10. Secondary Outcome: Change From Baseline to 6 Months Measurement of Pre-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at six months are included in the analysis
Time Frame: Baseline (Day 0) and 6 months after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 144 | 140 | 145 | 149
L | 0.14 [0.06 to 0.21] | 0.09 [0.01 to 0.16] | 0.10 [0.03 to 0.18] | 0.11 [0.04 to 0.18]

11. Secondary Outcome: Change From Baseline to 2 Weeks Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at two weeks are included in the analysis
Time Frame: Baseline (Day 0) and 2 weeks after Day 0
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 146 | 139 | 143 | 146
L | 0.06 [0.01 to 0.11] | 0.05 [-0.01 to 0.10] | 0.03 [-0.02 to 0.09] | 0.03 [-0.02 to 0.09]

12. Secondary Outcome: Change From Baseline to 1 Month Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at one month are included in the analysis
Time Frame: Baseline (Day 0) and 1 month after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 144 | 140 | 141 | 142
L | 0.06 [0.01 to 0.12] | 0.05 [0.00 to 0.11] | 0.03 [-0.03 to 0.09] | 0.03 [-0.03 to 0.08]

13. Secondary Outcome: Change From Baseline to 2 Months Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at two months are included in the analysis
Time Frame: Baseline (Day 0) and 2 months after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 142 | 138 | 141 | 142
L | 0.03 [-0.02 to 0.09] | 0.04 [-0.02 to 0.10] | 0.01 [-0.05 to 0.07] | 0.02 [-0.04 to 0.08]

14. Secondary Outcome: Change From Baseline to 3 Months Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at three months are included in the analysis
Time Frame: Baseline (Day 0) and 3 months after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 138 | 136 | 141 | 143
L | 0.04 [-0.02 to 0.10] | 0.04 [-0.02 to 0.10] | -0.00 [-0.06 to 0.06] | -0.01 [-0.07 to 0.05]

15. Secondary Outcome: Change From Baseline to 4 Months Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at four months are included in the analysis
Time Frame: Baseline (Day 0) and 4 months after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 141 | 136 | 141 | 141
L | 0.06 [-0.00 to 0.12] | 0.06 [0.00 to 0.13] | 0.03 [-0.03 to 0.10] | 0.03 [-0.03 to 0.10]

16. Secondary Outcome: Change From Baseline to 6 Months Measurement of Post-bronchodilator FEV1
Description: Only patients with both a non-missing value at baseline and visit at six months are included in the analysis
Time Frame: Baseline (Day 0) and 6 months after Day 0
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 139 | 136 | 142 | 145
L | 0.06 [0.01 to 0.12] | 0.02 [-0.03 to 0.08] | 0.04 [-0.02 to 0.10] | -0.01 [-0.07 to 0.05]

17. Secondary Outcome: Change From Baseline to Overall Mean of Treatment Period in ACQ-5 (Asthma Control Questionnaire, 5-item Version) Total Score
Description: The ACQ-5 is a validated questionnaire consisting of 5 items for the assessment of asthma symptom which are night symptom, morning symptom, limitation for the activities, shortness of breath, and wheeze. Each item is graded on a scale of 0-6 and the questions are equally weighted. The ACQ-5 score is the mean of the 5 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: Baseline (Day 0), Treatment Period (1,2,3,4, and 6 months)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale]
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 154 | 149 | 149 | 156
Units on a scale] | -0.68 [-0.83 to -0.52] | -0.66 [-0.82 to -0.51] | -0.64 [-0.80 to -0.48] | -0.70 [-0.86 to -0.55]

18. Secondary Outcome: Number of Patients Presenting Improvement From Baseline to End of Treatment Period in ACQ-5 (Asthma Control Questionnaire, 5-item Version)
Description: as for outcome 17
Time Frame: Baseline (Day 0) and 6 months after Day 0
Population: Full Analysis set
Measure: Number; unit: Participants with improvement
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 133 | 134 | 134 | 141
Participants with improvement | 72 | 88 | 73 | 69

19. Secondary Outcome: Change From Baseline to Overall Mean of Treatment Period in AQLQ(S) (Asthma Quality of Life Questionnaire Standardised Version) Overall Score
Description: The AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments in asthma. Patients are asked to score each item on a 7-point scale based on the experience of last 2 weeks. The overall AQLQ score is the mean response to all 32 questions. Therefore, the possible highest score (better) would be 7 and the lowest (worse) would be 1. Changes in scores of 0.5 to 1.0 are considered clinically meaningful; 1.0 to 1.5 as moderate and > 1.5 as marked clinically important differences for any individual domain or for the overall summary score.
Time Frame: Baseline (Day 0), Treatment Period (1,3, and 6 months)
Measure: Least Squares Mean (90% Confidence Interval); unit: Overall Score
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 152 | 145 | 145 | 153
Overall Score | 0.50 [0.36 to 0.65] | 0.46 [0.31 to 0.61] | 0.52 [0.37 to 0.67] | 0.52 [0.38 to 0.67]

20. Secondary Outcome: Number of Patients Presenting Improvement From Baseline to End of Treatment Period in AQLQ(S) (Asthma Quality of Life Questionnaire Standardised Version) Overall Score
Description: as for outcome 19
Time Frame: Baseline (Day 0) and 6 months after Day 0
Population: Full Analysis set
Measure: Number; unit: Participants with improvement
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 132 | 132 | 131 | 139
Participants with improvement | 62 | 68 | 69 | 62

21. Secondary Outcome: Change From Baseline to Treatment Period (Day 1 to Day 28) for Astma Symptom Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 1 to 28)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: Asthma symptom free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 160 | 153 | 156 | 159
Asthma symptom free days | -0.4 [-3.4 to 2.7] | 1.6 [-1.5 to 4.6] | 1.2 [-2.0 to 4.3] | 1.1 [-1.9 to 4.1]

22. Secondary Outcome: Change From Baseline to Treatment Period (Day 29 to Day 56) for Astma Symptom Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 29 to 56)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: symptom free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 158 | 148 | 152 | 155
symptom free days | 0.2 [-4.3 to 4.7] | 2.6 [-2.0 to 7.1] | 3.4 [-1.2 to 8.1] | 3.1 [-1.4 to 7.6]

23. Secondary Outcome: Change From Baseline to Treatment Period (Day 57 to Day 84) for Asthma Symptom Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 57 to 84)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: symptom free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 155 | 146 | 149 | 154
symptom free days | 1.4 [-3.4 to 6.3] | 4.3 [-0.6 to 9.3] | 3.0 [-2.1 to 8.0] | 4.0 [-0.9 to 8.9]

24. Secondary Outcome: Change From Baseline to Treatment Period (Day 85 to End of Treatment [6 Months]) for Asthma Symptom Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Day 85 to 6 months)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: symptom free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 152 | 145 | 148 | 151
symptom free days | 2.6 [-2.5 to 7.8] | 5.6 [0.5 to 10.7] | 3.9 [-1.3 to 9.2] | 4.4 [-0.7 to 9.5]

25. Secondary Outcome: Change From Baseline to Treatment Period (Day 1 to Day 28) for Asthma Control Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 1 to 28)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: asthma control days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 160 | 153 | 156 | 159
asthma control days | -1.1 [-3.9 to 1.6] | 1.7 [-1.1 to 4.6] | 1.2 [-1.7 to 4.1] | 0.9 [-1.8 to 3.7]

26. Secondary Outcome: Change From Baseline to Treatment Period (Day 29 to Day 56) for Asthma Control Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 29 to 56)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: asthma control days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 158 | 148 | 151 | 155
asthma control days | -0.1 [-4.2 to 4.0] | 3.5 [-0.7 to 7.7] | 2.7 [-4.2 to 4.0] | 2.8 [-1.4 to 6.9]

27. Secondary Outcome: Change From Baseline to Treatment Period (Day 57 to Day 84) for Asthma Control Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 57 to 84)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: asthma control days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 155 | 146 | 149 | 154
asthma control days | 0.9 [-3.8 to 5.6] | 4.7 [-0.0 to 9.4] | 3.2 [-1.6 to 8.1] | 2.9 [-1.8 to 7.6]

28. Secondary Outcome: Change From Baseline to Treatment Period (Day 85 to End of Treatment [6 Months]) for Asthma Control Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 85 to 6 months
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: asthma control days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 152 | 145 | 148 | 151
asthma control days | 1.4 [-3.4 to 6.2] | 5.7 [0.9 to 10.5] | 3.9 [-1.0 to 8.8] | 2.4 [-2.3 to 7.2]

29. Secondary Outcome: Change From Baseline to Treatment Period (Day 1 to Day 28) for Use of Rescue Medication Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 1 to 28)
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: rescue medication free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 160 | 153 | 156 | 159
rescue medication free days | 4.0 [-0.6 to 8.6] | 8.3 [3.6 to 13.0] | 6.8 [2.0 to 11.5] | 9.5 [4.9 to 14.1]

30. Secondary Outcome: Change From Baseline to Treatment Period (Day 29 to Day 56) for Use of Rescue Medication Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 29 to 56)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: rescue medication free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 158 | 148 | 150 | 155
rescue medication free days | 10.7 [4.6 to 16.8] | 17.6 [11.4 to 23.8] | 15.4 [9.1 to 21.8] | 16.4 [10.3 to 22.6]

31. Secondary Outcome: Change From Baseline to Treatment Period (Day 57 to Day 84) for Use of Rescue Medication Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 57 to 84)
Measure: Least Squares Mean (90% Confidence Interval); unit: rescue medication free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 155 | 146 | 147 | 153
rescue medication free days | 12.3 [5.7 to 18.9] | 19.2 [12.6 to 25.9] | 19.8 [13.0 to 26.6] | 18.7 [12.1 to 25.3]

32. Secondary Outcome: Change From Baseline to Treatment Period (Day 85 to End of Treatment [6 Months]) for Use of Rescue Medication Free Days
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 85 to 6 months)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: rescue medication free days
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 152 | 145 | 147 | 150
rescue medication free days | 15.8 [9.0 to 22.7] | 23.1 [16.2 to 29.9] | 21.2 [14.2 to 28.2] | 20.0 [13.2 to 26.8]

33. Secondary Outcome: Change From Baseline to Treatment Period (Day 1 to Day 28) for Night Time Awakenings Due to Asthma Symptoms
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Days 1 to 28)
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: night time awakenings
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 161 | 153 | 156 | 159
night time awakenings | -10.1 [-14.6 to -5.5] | -11.1 [-15.7 to -6.5] | -11.3 [-16.0 to -6.6] | -8.9 [-13.4 to -4.3]

34. Secondary Outcome: Change From Baseline to Treatment Period (Day 29 to Day 56) for Night Time Awakenings Due to Asthma Symptoms
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Day 29 to Day 56)
Population: Full Analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: night time awakenings
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 158 | 148 | 152 | 156
night time awakenings | -15.2 [-20.7 to -9.8] | -19.0 [-24.5 to -13.5] | -18.2 [-23.8 to -12.6] | -15.2 [-20.7 to -9.7]

35. Secondary Outcome: Change From Baseline to Treatment Period (Day 57 to Day 84) for Night Time Awakenings Due to Asthma Symptoms
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Day 57 to Day 84)
Population: full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: night time awakenings
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 155 | 146 | 149 | 154
night time awakenings | -17.6 [-23.2 to -11.9] | -19.8 [-25.5 to -14.0] | -22.1 [-27.9 to -16.2] | -16.7 [-22.4 to -11.0]

36. Secondary Outcome: Change From Baseline to Treatment Period (Day 85 to End of Treatment [6 Months]) for Night Time Awakenings Due to Asthma Symptoms
Time Frame: Baseline (last 14 days before randomization) and Treatment Period (Day 85 to 6 months)
Population: Full analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: night time awakenings
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 153 | 145 | 148 | 152
night time awakenings | -22.8 [-28.7 to -17.0] | -25.5 [-31.3 to -19.6] | -25.3 [-31.3 to -19.3] | -21.8 [-27.7 to -16.0]

37. Secondary Outcome: Number of Participants With Well Controlled Asthma Weeks at Baseline
Time Frame: Last 2 weeks before randomization
Measure: Number; unit: participants
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 160 | 153 | 156 | 159
participants
  0 Well-controlled asthma weeks Baseline | 154 | 152 | 150 | 152
  1 Well-controlled asthma weeks Baseline | 6 | 1 | 4 | 7
  2 Well-controlled asthma weeks Baseline | 0 | 0 | 2 | 0

38. Secondary Outcome: Number of Well Controlled Asthma Weeks During Treatment
Time Frame: Day 1to end of the 6 months treatment period
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: well controlled asthma weeks
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 162 | 156 | 160 | 158
well controlled asthma weeks | 1.7 (4.38) | 1.9 (4.78) | 2.4 (5.38) | 2.3 (5.27)

39. Secondary Outcome: Number of Participants With Uncontrolled Persistent Asthma Weeks at Baseline
Time Frame: Last 2 weeks before randomization
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 160 | 153 | 156 | 158
participants
  0 uncontrolled persistent asthma weeks | 23 | 18 | 26 | 27
  1 uncontrolled persistent asthma weeks | 40 | 39 | 34 | 36
  2 uncontrolled persistent asthma weeks | 97 | 96 | 96 | 95

40. Secondary Outcome: Number of Uncontrolled Persistent Asthma Weeks During Treatment
Time Frame: Day 1 to end of the 6 months treatment period
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: uncontrolled persistent asthma weeks
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 162 | 156 | 160 | 157
uncontrolled persistent asthma weeks | 11.0 (10.0) | 10.7 (10.02) | 10.4 (9.84) | 10.9 (9.89)

41. Secondary Outcome: Mean Plasma Concentration of AZD5069 at Day 7
Time Frame: Day 7
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/L)
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 159 | 147 | 144 | 0
(nmol/L) | 235.0 (1525.49) | 69.9 (717.83) | 25.4 (511.02) |

42. Secondary Outcome: Mean Plasma Concentration of AZD5069 at 1 Month
Time Frame: at 1 month
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/L)
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Number analyzed (Participants) | 148 | 135 | 139 | 0
(nmol/L) | 152.2 (11200.64) | 76.4 (788.17) | 25.8 (449.02) |

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | AZD5069 45 mg BID | AZD5069 15 mg BID | AZD5069 5 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 14/161 | 8/153 | 7/156 | 13/159
Other Adverse Events (participants affected / at risk) | 86/161 | 68/153 | 74/156 | 96/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5069 45 mg BID (N=161) | AZD5069 15 mg BID (N=153) | AZD5069 5 mg BID (N=156) | Placebo (N=159)
PNEUMONIA (Infections and infestations) | 3 | 1 | 0 | 2
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
SALMONELLOSIS (Infections and infestations) | 0 | 1 | 0 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 1
PERIPHERAL EMBOLISM (Vascular disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 3
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
BARRETTS OESOPHAGUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 0 | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PSEUDOHYPOPARATHYROIDISM (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5069 45 mg BID (N=161) | AZD5069 15 mg BID (N=153) | AZD5069 5 mg BID (N=156) | Placebo (N=159)
NASOPHARYNGITIS (Infections and infestations) | 18 | 13 | 18 | 31
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 4 | 4 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 3 | 2 | 3
DIARRHOEA (Gastrointestinal disorders) | 4 | 0 | 2 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
HEADACHE (Nervous system disorders) | 12 | 12 | 6 | 15
BRONCHITIS (Infections and infestations) | 7 | 6 | 1 | 10
PHARYNGITIS (Infections and infestations) | 3 | 4 | 5 | 5
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 3 | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2 | 6 | 3
INFLUENZA (Infections and infestations) | 3 | 3 | 4 | 3
PNEUMONIA (Infections and infestations) | 4 | 2 | 1 | 3
RHINITIS (Infections and infestations) | 2 | 4 | 1 | 0
SINUSITIS (Infections and infestations) | 3 | 1 | 3 | 5
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1 | 1 | 3
URINARY TRACT INFECTION (Infections and infestations) | 3 | 3 | 0 | 2
GASTROENTERITIS (Infections and infestations) | 1 | 2 | 1 | 2
Other (Infections and infestations) | 0 | 1 | 4 | 0
Other (Nervous system disorders) | 5 | 2 | 3 | 3
Other (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1 | 7
Other (Gastrointestinal disorders) | 8 | 4 | 1 | 7
Other (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5 | 5
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days